CLINICAL TRIAL: NCT06387264
Title: Efficacy and Safety of Medical Adhesive in the Treatment of Varicose Veins of the Lower Extremities: A Prospective, Multicenter, Randomized Controlled Study
Brief Title: Compont - Varicose Veins of the Lower Extremities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University First Hospital (Other); The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Liaocheng People's Hospital (Other); The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Zhang Xiaoming, Chief physician of Vascular Surgery, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022PHC032
Record Dates: First submitted 2024-04-16; First posted 2024-04-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Varicose Veins of Lower Limb
Keywords: Varicose Veins of Lower Limb; NBCA
MeSH Terms: interventions — Catheters

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical Adhesive treatment group (Experimental)
  Interventions: Device: Medical Adhesive
- Endovenous Radiofrequency Ablation Catheter (Active Comparator)
  Interventions: Device: ClosureFast Endovenous Radiofrequency Ablation(RFA) Catheter

INTERVENTIONS:
Device: Medical Adhesive — Medical Adhesive (produced by Beijing Compont Medical Devices Co., Ltd.) For varicose veins in the main saphenous vein, use 0.1 ml glue for every 3 cm of blood vessels.
  Arms: Medical Adhesive treatment group
Device: ClosureFast Endovenous Radiofrequency Ablation(RFA) Catheter — ClosureFast Endovenous Radiofrequency Ablation (RFA) Catheter (produced by America Medtronic Inc.) The ClosureFast catheter precisely heats a 7 cm vein segment in one 20-second interval.
  Arms: Endovenous Radiofrequency Ablation Catheter

SUMMARY:
The purpose of this clinical trial is to evaluate the effectiveness and safety of Medical Adhesive produced by Beijing Compont Medical Devices Co., Ltd. in the treatment of varicose veins in the lower extremities.

The main questions it aims to answer is: What medical problems do participants have when using tissue glue? Researchers will compare Medical Adhesive to ClosureFast Endovenous Radiofrequency Ablation (RFA) Catheter (produced by Medtronic Inc. to see if Medical Adhesive works to treat varicose veins in the lower extremities.

Participants will:

Treated with closed varicose veins of the lower extremity by Medical Adhesive or ClosureFast.

Return to the hospital at 1, 12, and 24 weeks postoperatively for Doppler ultrasound, and at 4, 12, 24 weeks postoperatively for venous scoring.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as great saphenous vein varices. (This operation only dealt with one side varicose veins of the lower extremities.)
* CEAP is graded C2-C6.
* Doppler ultrasound confirmed the patency of deep veins of lower limbs.
* Sign informed consent, voluntarily participate in the trial and follow up as required

Exclusion Criteria:

* A history of lower extremity deep vein thrombosis or pulmonary embolism
* Recurrent varicose veins
* The diameter of target lesion of the great saphenous vein less than 2 mm or more than 15 mm
* The great saphenous vein is severely distorted or tuberculated at the root
* Sepsis or septicemia
* Allergic to n-butyl cyanoacrylate
* The distance between the skin and the target vessel wall of the great saphenous vein less than 5 mm
* Severe cardiopulmonary disease, shock, coma or multiple organ failure
* Lactating or pregnant women
* Participated in other clinical trials within 1 month before surgery
* The researchers considered it unsuitable for inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Clinical success rate | 24 weeks after operation.
  At 24 weeks after surgery, Doppler ultrasound was used to check the closure of the target blood vessels.

SECONDARY OUTCOMES:
Technical success rate | Immediately after operation
  Immediately after operation, Doppler ultrasound was used to check the closure of the target blood vessels.
Target vascular closure rate at 12 weeks after operation. | 12 weeks after operation.
  At 12 weeks after surgery, Doppler ultrasound was used to check the closure of the target blood vessels.
Clinical signs | Screening period, 12 and 24 weeks after operation.
  The severity of the patient's clinical presentation was assessed according to the Clinical signs- etiologic classification- anatomic distribution- pathophysiologic dysfunction classification (CEAP classification) criteria.
  classification are as follows. C0: Without any visible or palpable signs of disease. C1: Telangiectasia or reticular veins C2: Varicose veins C2r: Recurrent varicose veins C3: Edema is present. C4: Changes in skin and subcutaneous tissue C4a: Pigmentation or eczema C4b: Lipodermatosclerosis or atrophie blanche C4c: Corona phlebectatica C5: Healed ulcers C6: Active ulcers C6r: Recurrent active venous ulcer
Venous Clinical Severity Score (VCSS) | Screening period, 4 weeks, 12 weeks and 24 weeks after operation.
  The VCSS score ranges from 0 to 30, with a larger value indicating approximately severe symptoms.
Aberdeen Varicose Vein Questionnaire (AVVQ) | Screening period, 4 weeks, 12 weeks and 24 weeks after operation.
  AVVQ scores range between 0 and 33, a higher score indicates a lower quality of life for patients.
Operation duration | Immediately after operation
Evaluation of product performance | within 24 hours after operation
  The researchers evaluated the operation performance of the product from the aspects of ease of operation and injection function, and divided the evaluation into three levels: satisfactory, general and unsatisfactory.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balint R, Farics A, Parti K, Vizsy L, Batorfi J, Menyhei G, Balint IB. Which endovenous ablation method does offer a better long-term technical success in the treatment of the incompetent great saphenous vein? Review. Vascular. 2016 Dec;24(6):649-657. doi: 10.1177/1708538116648035. Epub 2016 Apr 28. PMID 27126643
- [Background] Morrison N, Gibson K, McEnroe S, Goldman M, King T, Weiss R, Cher D, Jones A. Randomized trial comparing cyanoacrylate embolization and radiofrequency ablation for incompetent great saphenous veins (VeClose). J Vasc Surg. 2015 Apr;61(4):985-94. doi: 10.1016/j.jvs.2014.11.071. Epub 2015 Jan 31. PMID 25650040
- [Background] Morrison N, Gibson K, Vasquez M, Weiss R, Cher D, Madsen M, Jones A. VeClose trial 12-month outcomes of cyanoacrylate closure versus radiofrequency ablation for incompetent great saphenous veins. J Vasc Surg Venous Lymphat Disord. 2017 May;5(3):321-330. doi: 10.1016/j.jvsv.2016.12.005. Epub 2017 Mar 6. PMID 28411697
- [Background] Dimech AP, Cassar K. Efficacy of Cyanoacrylate Glue Ablation of Primary Truncal Varicose Veins Compared to Existing Endovenous Techniques: A Systematic Review of the Literature. Surg J (N Y). 2020 Jun 19;6(2):e77-e86. doi: 10.1055/s-0040-1708866. eCollection 2020 Apr. PMID 32577526
- [Background] Beteli CB, Rossi FH, de Almeida BL, Izukawa NM, Onofre Rossi CB, Gabriel SA, Kambara AM, de Moraes Rego Sousa AG, Thorpe P. Prospective, double-blind, randomized controlled trial comparing electrocoagulation and radiofrequency in the treatment of patients with great saphenous vein insufficiency and lower limb varicose veins. J Vasc Surg Venous Lymphat Disord. 2018 Mar;6(2):212-219. doi: 10.1016/j.jvsv.2017.09.010. Epub 2017 Dec 9. PMID 29229466
- [Background] Nordon IM, Hinchliffe RJ, Brar R, Moxey P, Black SA, Thompson MM, Loftus IM. A prospective double-blind randomized controlled trial of radiofrequency versus laser treatment of the great saphenous vein in patients with varicose veins. Ann Surg. 2011 Dec;254(6):876-81. doi: 10.1097/SLA.0b013e318230af5a. PMID 21934487